CLINICAL TRIAL: NCT01568515
Title: A Randomized Longitudinal Intervention Study to Assess Whether Electronic Messaging Can Increase HPV Vaccine Utilization and Adherence Among College Students in Eastern North Carolina.
Brief Title: Electronic Messaging to Increase Human Papillomavirus Vaccine Utilization and Adherence Among College Students
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dr. Alice Richman, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MISP-39631
Record Dates: First submitted 2012-03-22; First posted 2012-04-02 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Patient Compliance; Health Knowledge, Attitudes, Practice
Keywords: HPV vaccine; Vaccine adherence; Vaccine utilization; Electronic Messaging
MeSH Terms: conditions — Patient Compliance; Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic Messages (Experimental): Intervention group participants received electronic (text and/or email) reminder messages coupled with health educational messages about HPV and HPV vaccine across 7 months
  Interventions: Procedure: Electronic Message
- Standard of Care (No Intervention): Control group participants received standard of care at the student health center which included a card with their next appointment written on it.

INTERVENTIONS:
Procedure: Electronic Message — Students enrolled in the intervention group received 7 electronic contacts over a 7-month period. Specifically, participants received 4 electronic education messages, 2 electronic reminder/education messages, as well as 1 baseline and 1 final assessment contacts. Up to 4 reminder contacts were used if surveys were not completed for both intervention and control group participants. Control group participants will receive 2 contacts throughout the study, 1 at baseline and 1 at their final assessment. Up to 4 reminder contacts were used if surveys were not completed. Intervention & control groups were compared longitudinally for 7 months on the differences in HPV vaccine utilization and adherence, knowledge and attitudes about HPV, and the HPV vaccine (parallel design).
  Arms: Electronic Messages

SUMMARY:
Introduction: Although vaccination against HPV and subsequent HPV-related cancers is a significant breakthrough, uptake is low. We sought to understand whether a low-cost intervention of electronic (text and/or email) appointment reminders coupled with electronic health educational messaging about HPV and the HPV vaccine could increase HPV vaccine uptake and knowledge among college students.

Methods: Study participants included both female and male English speaking students between the ages of 18-26 who attended a large university in North Carolina. Students were randomized to the intervention or control group. Intervention group participants received the electronic messaging while the control group received standard of care at the student health center across a 7-month study period. Baseline and follow-up survey data was collected. Main outcome measures were completion of HPV-2 and HPV-3 and HPV and HPV vaccine knowledge. Study recruitment ran from August 2011 to December 2013.

Results: Completion rates for the intervention and control group were similar for HPV-2 (53% vs. 52%) and HPV-3 (34% vs. 32%), respectively. The mean knowledge score at follow-up for intervention group participants (n=44, mean knowledge score = 93%, SD = 0.08) was significantly higher (p=0.01) than the mean knowledge score at baseline (n=44, mean knowledge score = 87%, SD = 0.11). No significant changes in knowledge from baseline to follow-up were found for control group participants. The single most important predictor of HPV vaccine uptake overall was female gender where female participants were 2.35 times [confidence interval (CI) 1.17-4.69] as likely to complete the series as compared to male participants.

Conclusion: In this sample of college students, the electronic messaging intervention increased knowledge but not uptake. More randomized controlled trials on the efficacy of HPV vaccine electronic reminder interventions for catch-up age populations for both females and males are needed.

DETAILED DESCRIPTION:
Oncogenic types of human papillomavirus (HPV) infection can cause cervical cancer, with HPV types 16 and 18 causing roughly 70% of cervical cancers worldwide.1 Persistent HPV infection has also been linked to vaginal and vulvar cancer in women, penile cancer in men, as well as oral pharyngeal cancer, anal cancer, and genital warts in both sexes.2-4 There are two safe and effective vaccines which protect against HPV types 16 and 18 and one of the two vaccines (HPV4) also protects against two additional HPV types that account for 90% of the cases of genital warts.5 Because HPV vaccination provides maximum protection if administered prior to sexual debut, HPV4 guidelines recommend administration to males and females ages 11 and 12, with catch-up vaccination up to age 26, for the prevention of cervical and anal cancers as well as for the prevention of genital warts.1,5-8 Although vaccination against HPV-related cancers is a significant breakthrough, uptake is low. The National Immunization Survey-Teen (NIS-teen) estimated that in 2013, HPV vaccination coverage for 13-17 year-old females was 37.6%, while for males in the same age group coverage was 13.9%. Additionally, coverage for 13-17 year-old females dropped slightly between 2011 and 2012.9 Although vaccination coverage for teens has been increasing over time overall, these rates are far from meeting the Healthy People 2020 goal of 80% of 13-15 year old females being fully vaccinated against HPV by 2020. In addition to teens, it has been shown that there is a benefit to providing HPV vaccines to young adults, even those who have already been sexually active. However, an NIS-adult study showed that only 10-12% of 18-26 year-old women are completing the HPV vaccine series.10 Additionally, studies have found significantly lower completion rates among African Americans.9,11-12 This is problematic given that African American women demonstrate a mortality rate from cervical cancer that is twice that of Caucasian women.13 It has also been suggested that lack of knowledge may be a barrier to vaccine adherence14 and that educational interventions may increase adherence among 18-26 year-old women.12 Given the importance of immunizing young adults for the prevention of cancer and given the low uptake of HPV vaccines in this group, it is important to develop and evaluate strategies to increase use and adherence among this population. We sought to understand whether a low-cost intervention of electronic (text and/or email) appointment reminders coupled with electronic health educational messaging about HPV and the HPV vaccine could increase HPV vaccine utilization, adherence, and knowledge among college students (both female and male) attending a large university in eastern North Carolina. Although we only found one peer-reviewed study that assessed text and email electronic HPV reminders primarily among adolescents, we found a few other studies that assessed mail and telephone HPV vaccination reminders among adolescents. All of these studies found vaccination reminders to be effective in increasing adherence among adolescents and/or young adults.15-17 Hard copy and electronic messaging reminders have also proven to be effective when coupled with other prevention strategies such as immunizations for influenza and pneumococcal pneumonia as well as screening for colon, breast, and cervical cancer in adults.18 We found no literature that tested electronic HPV vaccine interventions among a college population.

Our primary hypothesis was that students who receive the intervention would be more compliant in their uptake of the second (HPV-2) and third (HPV-3) doses of the vaccine as compared to the control group. Secondarily, we further hypothesized that students that receive the intervention will demonstrate higher knowledge about HPV and the HPV vaccine as compared to the control group and that African American students and younger students (defined as 18-19 years of age) would be less compliant as compared to Caucasian and older students (defined as students 20 and older), as demonstrated in the literature. Lastly, we sought to describe satisfaction of health messages and reminders among those that received it.

ELIGIBILITY:
Inclusion Criteria:

* Male & Female Students enrolled at East Carolina University (ECU)

Exclusion Criteria:

* Non-English speaking students
* Students under the age of 18 or over 26
* Individuals not enrolled at ECU

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 283 (Actual)
Dates: Start 2011-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Increase in HPV vaccine uptake among intervention group participants. | One year
  To determine if electronic reminders coupled with electronic educational messaging can increase HPV vaccine use and adherence among college students in eastern North Carolina.

SECONDARY OUTCOMES:
Increase knowledge of HPV and HPV vaccine among intervention group participants | One year
  To measure whether electronic health educational messaging increases HPV and HPV vaccine knowledge among college students in eastern North Carolina.
Compliance rates among Race/ethnicity and other socio-demographic characteristics. | One year
  We hypothesize that African American students and younger students (defined as 18-19 years of age) will be less compliant as compared to Caucasian and older students (defined as students 20 and older) as demonstrated in the literature. Items measuring race/ethnicity and socio-demographic variables will be included on baseline and follow-up surveys. We will assess whether these variables predict vaccine adherence among study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Alice R Richman, PhD, Principal Investigator — East Carolina University

REFERENCES:
- [Background] Saslow D, Solomon D, Lawson HW, Killackey M, Kulasingam SL, Cain J, Garcia FA, Moriarty AT, Waxman AG, Wilbur DC, Wentzensen N, Downs LS Jr, Spitzer M, Moscicki AB, Franco EL, Stoler MH, Schiffman M, Castle PE, Myers ER; American Cancer Society; American Society for Colposcopy and Cervical Pathology; American Society for Clinical Pathology. American Cancer Society, American Society for Colposcopy and Cervical Pathology, and American Society for Clinical Pathology screening guidelines for the prevention and early detection of cervical cancer. Am J Clin Pathol. 2012 Apr;137(4):516-42. doi: 10.1309/AJCPTGD94EVRSJCG. PMID 22431528
- [Background] Hoots BE, Palefsky JM, Pimenta JM, Smith JS. Human papillomavirus type distribution in anal cancer and anal intraepithelial lesions. Int J Cancer. 2009 May 15;124(10):2375-83. doi: 10.1002/ijc.24215. PMID 19189402
- [Background] Kreimer AR, Clifford GM, Boyle P, Franceschi S. Human papillomavirus types in head and neck squamous cell carcinomas worldwide: a systematic review. Cancer Epidemiol Biomarkers Prev. 2005 Feb;14(2):467-75. doi: 10.1158/1055-9965.EPI-04-0551. PMID 15734974
- [Background] Gillison ML, Chaturvedi AK, Lowy DR. HPV prophylactic vaccines and the potential prevention of noncervical cancers in both men and women. Cancer. 2008 Nov 15;113(10 Suppl):3036-46. doi: 10.1002/cncr.23764. PMID 18980286
- [Background] Centers for Disease Control and Prevention (CDC). FDA licensure of bivalent human papillomavirus vaccine (HPV2, Cervarix) for use in females and updated HPV vaccination recommendations from the Advisory Committee on Immunization Practices (ACIP). MMWR Morb Mortal Wkly Rep. 2010 May 28;59(20):626-9. PMID 20508593
- [Background] Jain N, Euler GL, Shefer A, Lu P, Yankey D, Markowitz L. Human papillomavirus (HPV) awareness and vaccination initiation among women in the United States, National Immunization Survey-Adult 2007. Prev Med. 2009 May;48(5):426-31. doi: 10.1016/j.ypmed.2008.11.010. Epub 2008 Dec 6. PMID 19100762
- [Background] Elam-Evans LD, Yankey D, Jeyarajah J, Singleton JA, Curtis RC, MacNeil J, Hariri S; Immunization Services Division, National Center for Immunization and Respiratory Diseases; Centers for Disease Control and Prevention (CDC). National, regional, state, and selected local area vaccination coverage among adolescents aged 13-17 years--United States, 2013. MMWR Morb Mortal Wkly Rep. 2014 Jul 25;63(29):625-33. PMID 25055186
- [Background] Widdice LE, Bernstein DI, Leonard AC, Marsolo KA, Kahn JA. Adherence to the HPV vaccine dosing intervals and factors associated with completion of 3 doses. Pediatrics. 2011 Jan;127(1):77-84. doi: 10.1542/peds.2010-0812. Epub 2010 Dec 13. PMID 21149425
- [Background] Kester LM, Shedd-Steele RB, Dotson-Roberts CA, Smith J, Zimet GD. The effects of a brief educational intervention on human papillomavirus knowledge and intention to initiate HPV vaccination in 18-26 year old young adults. Gynecol Oncol. 2014 Mar;132 Suppl 1:S9-12. doi: 10.1016/j.ygyno.2013.12.033. Epub 2013 Dec 31. PMID 24384459
- [Background] American Cancer Society (ACS). Cancer Facts & Figures 2014.